CLINICAL TRIAL: NCT03673046
Title: Smartphone Cognitive Behavioral Therapy for Body Dysmorphic Disorder: A Randomized, Waitlist-control Trial
Brief Title: Waitlist-Control Trial of Smartphone Cognitive Behavioral Therapy (CBT) for Body Dysmorphic Disorder (BDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Koa Health B.V. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000293_B; NCT04034693 (obsolete NCT alias)
Record Dates: First submitted 2018-09-11; First posted 2018-09-17 (Actual); Results first posted 2022-09-14 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Body Dysmorphic Disorder
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD) (Experimental): 12-week Smartphone-delivered CBT for BDD.
  Interventions: Device: Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD)
- 12 Week Waitlist Control (Other): 12 week waitlist control. (Note: participants will be crossed over to 12-week Smartphone-delivered CBT for BDD following the 12-week waitlist control).
  Interventions: Device: Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD)

INTERVENTIONS:
Device: Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD) — 12-week Smartphone-delivered CBT for BDD. In-person cognitive behavioral therapy (CBT) is an empirically supported treatment for BDD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.

SUMMARY:
The investigators are testing the efficacy of Smartphone-delivered cognitive behavioral therapy (CBT) treatment for body dysmorphic disorder (BDD). The investigators hypothesize that participants receiving app-CBT will have greater improvement in body dysmorphic disorder symptom severity than those in the waitlist condition at treatment endpoint (week 12).

DETAILED DESCRIPTION:
The primary aim of this study is to test the efficacy of a Smartphone-based cognitive behavioral therapy (CBT) treatment for adults with body dysmorphic disorder (BDD) recruited nationally. In a prior study (Clinical Trials Identifier # NCT03221738), the investigators developed and pilot-tested the feasibility, acceptability, and preliminary efficacy of a CBT for BDD app in an open pilot trial. The investigators are now further testing these outcomes in a randomized controlled trial. Eligible subjects (N= 64) will be randomly assigned to 12-weeks of Smartphone-delivered CBT for BDD either immediately, or after a 12-week long waiting period (50/50 chance).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current diagnosis of primary body dysmorphic disorder (BDD), based on a clinical structured diagnostic interview
* currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment (Participants taking psychotropic medication must have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period)
* Past participation in 4+ sessions of cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD)
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation as indicated by clinical judgment and/or a score >2 on the suicidal ideation subscale of the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Current severe comorbid major depression, as indicated by clinical judgment and/or a Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR) total score ≥ 21
* Concurrent psychological treatment
* Does not own a supported Smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Weingarden H, Garriga Calleja R, Greenberg JL, Snorrason I, Matic A, Quist R, Harrison O, Hoeppner SS, Wilhelm S. Characterizing observed and effective behavioral engagement with smartphone cognitive behavioral therapy for body dysmorphic disorder: A methods roadmap and use case. Internet Interv. 2023 Mar 16;32:100615. doi: 10.1016/j.invent.2023.100615. eCollection 2023 Apr. PMID 36969390

RESULTS

PARTICIPANT FLOW:
Groups:
- Smartphone-delivered Cognitive Behavioral Therapy (CBT) for Body Dysmorphic Disorder (BDD): 12-week Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD). In-person CBT is an empirically supported treatment for BDD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.
- Waitlist Control: 12-week waitlist control. (Note: participants will be crossed over to 12-week Smartphone-delivered cognitive behavioral therapy (CBT) for body dysmorphic disorder (BDD) following the 12-week waitlist control).
Period: Overall Study
Arm/Group | Smartphone-delivered Cognitive Behavioral Therapy (CBT) for Body Dysmorphic Disorder (BDD) | Waitlist Control
Started | 40 | 40
Completed | 31 | 37
Not Completed | 9 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone-delivered Cognitive Behavioral Therapy (CBT) for Body Dysmorphic Disorder (BDD) | Waitlist Control | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (9.9) | 26.2 (9.5) | 27.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 30 | 67
  Male | 3 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 36 | 34 | 70
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 22 | 55
  Asian | 4 | 8 | 12
  Black / African American | 0 | 2 | 2
  More than one race | 3 | 5 | 8
  Other | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Education [Count of Participants; unit: Participants]
  Some high school | 0 | 1 | 1
  High school diploma / General Educational Development (GED) diploma | 8 | 5 | 13
  Some college | 9 | 7 | 16
  2-year degree / certificate | 2 | 4 | 6
  College graduate | 11 | 11 | 22
  Some post-graduate / professional | 2 | 3 | 5
  Post-graduate / professional degree | 8 | 9 | 17
Marital status [Count of Participants; unit: Participants]
  Single / never married | 30 | 28 | 58
  Married (including Common Law) | 7 | 7 | 14
  Living with partner | 2 | 2 | 4
  Divorced / separated | 1 | 3 | 4
Duration of body dysmorphic disorder (BDD), years [Mean (Standard Deviation); unit: years] — Population: Two participants in the immediate smartphone CBT group had missing data for age of onset of BDD.
  years
    number analyzed (Participants) | 38 | 40 | 78
    (all) | 14.0 (9.9) | 12.6 (11.6) | 13.3 (10.7)
Number of body parts of concern, mean (standard deviation (SD)) [Mean (Standard Deviation); unit: Body parts/participant] — Participants used a checklist to identify all body parts of concern to them. The number of body parts checked by each participant were summed.
  Body parts/participant | 11.2 (6.3) | 11.1 (6.4) | 11.1 (6.3)
Delusional BDD [Count of Participants; unit: Participants] — Delusional beliefs about body dysmorphic disorder were assessed via the Brown Assessment of Beliefs Scale (BABS). Participants were deemed to be delusional if they had a BABS total score of 18 out of a possible total score of 24 in combination with a score of 4 on the first item (conviction).
  Participants | 4 | 4 | 8
Number of current comorbid MINI diagnoses [Count of Participants; unit: Participants] — The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a short structured diagnostic interview for psychiatric disorders included in the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V) and the International Classification of Diseases 10th Revision (ICD-10). Trained clinicians administered the diagnostic interview over approximately 15 minutes to identify whether participants met diagnostic criteria for relatively common (e.g., major depressive disorder) or related (e.g., eating disorders) current and past psychiatric disorders.
  Participants
    None | 13 | 14 | 27
    1 | 14 | 14 | 28
    2 | 8 | 8 | 16
    3 or more | 5 | 4 | 9
Enrolled after COVID-19 pandemic started [Count of Participants; unit: Participants] | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Difference in BDD Severity (BDD-YBOCS) at the End of Treatment/Waitlist Period.
Description: The BDD Yale-Brown Obsessive Compulsive Scale (BDD-YBOCS) is the gold-standard, semi-structured clinician-administered assessment of BDD severity. It contains 12 items ranging from 0 to 4, which are summed to generate a total score (range = 0 to 48). Higher scores indicate more severe BDD symptoms. The BDD-YBOCS
Time Frame: Week 0, Week 6, and Week 12
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Smartphone-delivered CBT for BDD: 12-week Smartphone-delivered CBT for BDD. In-person cognitive behavioral therapy (CBT) is an empirically supported treatment for BDD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.
- Waitlist Control: 12-week waitlist control. (Note: participants will be crossed over to 12-week Smartphone-delivered CBT for BDD following the 12-week waitlist control).
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
Number analyzed (Participants) | 40 | 40
score on a scale
  Week 0 | 29.85 (4.02) | 30.85 (4.82)
  Week 6: number analyzed (Participants) | 35 | 38
  Week 6 | 23.77 (6.93) | 27.13 (6.03)
  Week 12: number analyzed (Participants) | 31 | 37
  Week 12 | 16.81 (7.47) | 26.70 (6.24)
Statistical Analysis 1: Comparison: Smartphone-delivered CBT for BDD vs Waitlist Control; Null hypothesis: there is no significant difference in BDD-YBOCS total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p < .0001, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was the pre-specified primary endpoint comparison. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with a compound symmetry with heterogeneous variance covariance matrix; Mean Difference (Final Values) = -10.1255, 95% CI 2-sided [-13.2532 to -6.9978], Standard Error of Mean 1.5705 — The effect is presented as the Smartphone-delivered CBT for BDD group outcome compared to the 12-eeek waitlist control group outcome at the trial end-point (week 12)

2. Secondary Outcome: Difference in Depression at the End of Treatment/Waitlist Period
Description: The self-report Quick Inventory of Depressive Symptomatology (QIDS-SR) is a measure of depressive symptoms consisting of 16 scale items with responses ranging from 0 to 3, including one suicide item (item #12). Total scores have a range from 0 to 27 with higher scores indicating greater depression severity. The measure is a well-validated, sensitive measure of symptom severity in depression.
Time Frame: Week 0, Week 6, and Week 12
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
Number analyzed (Participants) | 40 | 40
score on a scale
  Week 0 | 11.13 (4.37) | 11.43 (3.96)
  Week 6: number analyzed (Participants) | 34 | 36
  Week 6 | 10.15 (4.77) | 10.08 (4.74)
  Week 12: number analyzed (Participants) | 28 | 36
  Week 12 | 7.11 (4.51) | 10.31 (4.17)
Statistical Analysis 1: Comparison: Smartphone-delivered CBT for BDD vs Waitlist Control; Null hypothesis: there is no significant difference in QIDS-SR total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p = 0.0023, Mixed Models Analysis — The p-value was not adjusted for multiple comparisons because this was a pre-specified secondary endpoint comparison. The a priori threshold for statistical significance was alpha=.05; Repeated measures were modeled with an auto-correlation with heterogeneous variance (ARH(1)) covariance matrix; Mean Difference (Final Values) = -3.2648, 95% CI 2-sided [-5.3275 to -1.2022], Standard Error of Mean 1.0346 — The effect is presented as the Smartphone-delivered CBT for BDD group outcome compared to the 12-week waitlist control group outcome at the trial end-point (week 12)

3. Secondary Outcome: Difference in Delusionality at the End of Treatment/Waitlist Period
Description: Delusionality was assessed using the Brown Assessment of Beliefs Scale (BABS). The BABS is a semi-structured, clinician-administered interview that assesses delusional thinking related to one's appearance concerns. It contains 7 items ranging from 0-4; the first six items are summed to generate a total score (range: 0-24). Higher scores indicate greater delusionality.
Time Frame: Week 0, Week 6, and Week 12
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
Number analyzed (Participants) | 40 | 40
score on a scale
  Week 0 | 15.10 (3.25) | 14.45 (3.43)
  Week 6: number analyzed (Participants) | 35 | 38
  Week 6 | 12.26 (5.25) | 13.50 (4.75)
  Week 12: number analyzed (Participants) | 30 | 37
  Week 12 | 8.30 (4.98) | 13.22 (4.88)
Statistical Analysis 1: Comparison: Smartphone-delivered CBT for BDD vs Waitlist Control; Null hypothesis: there is no significant difference in BABS total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p < .0001, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Repeated measures were modeled with a compound symmetry with heterogeneous variance covariance matrix; Mean Difference (Final Values) = -4.8412, 95% CI 2-sided [-7.0698 to -2.6126], Standard Error of Mean 1.1195 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Difference in Functional Impairment at the End of Treatment/Waitlist Period
Description: Functional impairment was measured using the Sheehan Disability Scale (SDS). The SDS is a self-rated, 3-item questionnaire that uses a Likert scale from 0 (not at all) to 10 (extremely) to assess impairment in occupational, social, and family domains. The 3 items are summed for a total score (range: 0-30), where higher scores indicate greater functional impairment.
Time Frame: Week 0, Week 6, and Week 12
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
Number analyzed (Participants) | 40 | 40
score on a scale
  Week 0 | 15.95 (6.56) | 17.08 (6.76)
  Week 6: number analyzed (Participants) | 34 | 37
  Week 6 | 11.09 (6.36) | 13.22 (7.21)
  Week 12: number analyzed (Participants) | 28 | 37
  Week 12 | 7.64 (6.78) | 13.49 (7.31)
Statistical Analysis 1: Comparison: Smartphone-delivered CBT for BDD vs Waitlist Control; Null hypothesis: there is no significant difference in SDS total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p = .0008, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Repeated measures were modeled with an auto-correlation with heterogeneous variance (ARH(1)) covariance matrix; Mean Difference (Final Values) = -5.8847, 95% CI 2-sided [-9.2237 to -2.5458], Standard Error of Mean 1.6760 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Difference in Quality of Life at the End of Treatment/Waitlist Period
Description: Quality of life was assessed using The Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). The Q-LES-Q-SF is a 16-item self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100), with higher scores indicating greater quality of life.
Time Frame: Week 0, Week 6, and Week 12
Population: Data was analyzed in an intent to treat analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
Number analyzed (Participants) | 40 | 40
score on a scale
  Week 0 | 52.72 (16.27) | 48.35 (10.19)
  Week 6: number analyzed (Participants) | 34 | 37
  Week 6 | 53.99 (16.42) | 52.12 (12.25)
  Week 12: number analyzed (Participants) | 28 | 37
  Week 12 | 66.45 (16.45) | 55.20 (12.40)
Statistical Analysis 1: Comparison: Smartphone-delivered CBT for BDD vs Waitlist Control; Null hypothesis: there is no significant difference in Q-LESQ-SF total scores between the treatment groups at endpoint (week 12); Test type: Superiority; p = .0011, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Repeated measures were modeled with a compound symmetry with heterogeneous variance covariance matrix; Mean Difference (Final Values) = 11.7529, 95% CI 2-sided [4.8630 to 18.6428], Standard Error of Mean 3.4553 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected every 6 weeks after the baseline visit, during the mid-treatment assessment visit (week 6) and the post-treatment visit (week 12). At these assessments, participants were probed for adverse events that occurred since the last adverse event assessment (usually 6 weeks prior).
Description: Participants were asked 4 questions about: (1) any major physical health problems or major physical injuries; (2) seeing a physical health or mental health provider for any reason; (3) any hospitalizations; or (4) any other major problems or concerns, all pertaining to the time since they were assessed last. Any "yes" resulted in a full event report. All serious adverse events are reported. Of non-serious events, only those affecting >5% in either treatment group are reported.
Arm/Group | Smartphone-delivered CBT for BDD | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 19/40 | 11/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Smartphone-delivered CBT for BDD (N=40) | Waitlist Control (N=40)
Increased anxiety or depression (Psychiatric disorders) | 5 | 1
Suicidal ideation worsening (Psychiatric disorders) | 5 | 1
Allergies, allergic reactions (Immune system disorders) | 3 | 2
Injuries and accidents (Injury, poisoning and procedural complications) | 3 | 1 — Shoulder/neck injuries, car accident, broken finger
Procedural complications (Injury, poisoning and procedural complications) | 0 | 2
Migraine (Nervous system disorders) | 2 | 0
Endometriosis (Reproductive system and breast disorders) | 2 | 0
Medical procedure (Surgical and medical procedures) | 2 | 1
Other (Psychiatric disorders) | 0 | 3 — panic attack, jaw pain, BDD symptom worsening

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT03673046/Prot_SAP_001.pdf